CLINICAL TRIAL: NCT05690945
Title: A Randomized, Double-blind, Multicenter Phase 3 Clinical Study to Evaluate the Efficacy and Safety of QL1706 in Combination With Chemotherapy in First-line PD-L1 Negative, Locally Advanced or Metastatic Non-small Cell Lung Cancer Patients
Brief Title: A Study of QL1706 in Combination With Chemotherapy in PD-L1-Negative Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QL1706-303
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1706+chemotherapy (Experimental): Participants with locally advanced or metastatic NSCLC patients who are PD-L1 negative will receive QL1706, paclitaxel/pemetrexed and carboplatin by intravenous (IV) injection on Day 1 of each 21-day cycle for 4 cycles in the induction treatment. In the maintenance phase, participants will be treated with QL1706 or QL1706 combined with pemetrexed.
  Interventions: Drug: QL1706
- Tiselizumab+chemotherapy (Active Comparator): Participants with locally advanced or metastatic NSCLC patients who are PD-L1 negative will receive tiselizumab, paclitaxel/pemetrexed and carboplatin by intravenous (IV) injection on Day 1 of each 21-day cycle for 4 cycles in the induction treatment. In the maintenance phase, participants will be treated with tiselizumab or tiselizumab combined with pemetrexed.
  Interventions: Drug: Tilesizumab

INTERVENTIONS:
Drug: QL1706 — QL1706 will be administered by IV infusion at 5mg/kg on Day 1 of each 21-day cycle until unacceptabletoxicity or loss of clinical benefit.
  Other Names: PSB205
  Arms: QL1706+chemotherapy
Drug: Tilesizumab — Tilesizumab will be administered by IV infusion at 200mg on Day 1 of each 21-day cycle until unacceptabletoxicity or loss of clinical benefit.
  Other Names: BGB-108
  Arms: Tiselizumab+chemotherapy

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of QL1706 combined with platinum-based chemotherapy versus tislelizumab combined with platinum-based chemotherapy in PD-L1 negative, locally advanced or metastatic Non-small Cell Lung Cancer Patients. The subjects were randomly divided into two groups according to 1:1, with about 304 subjects in the experimental group and the control group.

DETAILED DESCRIPTION:
This study was a randomized, double-blind, active-controlled, multicenter Phase 3 clinical study. The study is designed to evaluate the efficacy and safety of QL1706 in combination with chemotherapy or commercial PD1 in combination with chemotherapy in locally advanced or metastatic NSCLC patients who are PD-L1 negative.608 patients would be enrolled . Subjects will be assigned randomly in a 1:1 ratio to experimental group and control group. Subjects will be stratified by pathological type: squamous cell carcinoma versus non-squamous cell carcinoma; brain metastasis: present versus absent; gender: male versus female. After randomization, subjects will be treated according to the randomization results.

ELIGIBILITY:
Inclusion Criteria:

1. Be≥18 to ≤ 75 years of age at enrollment, male or female.
2. Histologically or cytologically confirmed locally advanced (Stage IIIB/IIIC) that not amenable to complete surgical resection and not amenable to radical concurrent/sequential chemoradiation or metastatic (Stage IV) NSCLC (American Joint Committee on Cancer [AJCC] 8th edition).
3. No EGFR sensitive mutations or ALK gene translocation alterations.
4. Capable of providing fresh or archived 2 years' tissue samples collected at post-diagnosis or non-radiation sites at diagnosis for central laboratory PD-L1 testing with TPS < 1% .
5. Have a life expectancy of at least 3 months.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. No prior systemic therapy for advanced or metastatic NSCLC was received.

Exclusion Criteria:

1. Previous treatment with immune checkpoint inhibitors (PD-1/PD-L1 drugs or drugs acting on another T cell receptor (e.g., CTLA-4 etc.), as well as immune checkpoint agonistic antibodies (e.g., anti ICOS , CD40 , CD137 , GITR , OX40 antibodies, etc.), and immune cell therapy.
2. Patients who have received systemic corticosteroids or other immunosuppressive drugs within 2 weeks prior to the first dose.
3. Presence or history of any active autoimmune disease, including, but not limited to: autoimmune hepatitis, interstitial pneumonia, pulmonary fibrosis, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism.
4. Pulmonary radiation therapy > 30 Gy within 6 months prior to first dose;
5. Palliative radiotherapy completed 7 days prior to first dose.
6. Known or symptomatic active central nervous system (CNS) metastases or carcinomatous meningitis during screening.
7. Clinically significant cardiovascular or cerebrovascular disease

   -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
OS | From date of randomization until the date of death from any cause, which ever came first, assessed up to 2 years
  Overall Survival (OS) in the ITT population determined by the investigator

SECONDARY OUTCOMES:
ORR | First administration until disease progression or death, which ever occurs first (up to approximately 24 months)
  Objective Response Rate assessed by investigator according to RECIST v1.1 criteria
DOR | First administration until disease progression or death, which ever occurs first (up to approximately 24 months)
  Duration of Response assessed by investigator according to RECIST v1.1 criteria
DCR | First administration until disease progression or death, which ever occurs first (up to approximately 24 months)
  Disease Control Rate assessed by investigator according to RECIST v1.1 criteria
PFS | Informed consent until disease progression or death, which ever occurs first (up to approximately 2 years)
  Progression Free Survival in the intent to treat (ITT) population, as determined by the investigator according to RECIST v1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Professor, Principal Investigator — Sun Yat-sen Univeisity Cancer Center
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China